CLINICAL TRIAL: NCT05059652
Title: Effects of Ischemic Preconditioning on Conditioned Pain Modulation and Heart Rate Variability in Women With Knee Osteoarthritis: Placebo-Controlled Randomized Clinical Trial
Brief Title: Effects of Ischemic Preconditioning on Conditioned Pain Modulation and Heart Rate Variability in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Principal Investigator, Paulista University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5543/2021
Record Dates: First submitted 2021-08-30; First posted 2021-09-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Preconditioning
Keywords: ischemic preconditioning; therapeutic occlusion; conditioned pain modulation; heart rate variability; autonomic nervous system; osteoarthritis; chronic pain
MeSH Terms: conditions — Osteoarthritis; Chronic Pain | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic Preconditioning (n= 22) (Experimental): The IPC protocol will be applied in the proximal region of the thigh of the limb with knee osteoarthritis and if both knees are affected, it will be applied to the knee with the greatest complaint of pain.
  Participants will be relaxed and comfortably seated. The same cuff used to determine the total occlusion pressure (TOP) will be used and the protocol will consist of four cycles of total ischemia (according to the TOP value determined individually) of five minutes, followed immediately by four cycles of five minutes of vascular reperfusion (0 mmHg ), totaling 40 minutes.
  Interventions: Device: Ischemic Preconditioning
- Placebo (n= 22) (Placebo Comparator): The placebo protocol will be performed on the lower limb with knee osteoarthritis and if both knees are affected, it will be applied to the knee with the greatest complaint of pain. Participants will perform a protocol similar to the IPC, but during the four cycles of five minutes of occlusion, the cuffs will only be inflated with 10mmHg so as not to cause arterial or venous occlusion, alternating with four cycles of five minutes of reperfusion (0 mmHg).
  Interventions: Device: Ischemic Preconditioning

INTERVENTIONS:
Device: Ischemic Preconditioning — The Ischemic Preconditioning (IPC) is characterized by the application of brief periods of circulatory occlusion (ischemia) and reperfusion of a limb in the minutes to hours that precede the exercise through the insufflations and deflations of a pressure cuff.

SUMMARY:
Introduction: Musculoskeletal disorders have affected approximately 1.3 billion people worldwide. Evidence shows that chronic diseases and musculoskeletal conditions often occur together, and among them it is estimated that more than 240 million people worldwide have symptomatic osteoarthritis (OA) and activity limitation, which is a major contributor to chronic pain and changes central in pain processing. It is known that physical exercise (active approach to treatment) and manual therapy (passive approach) are capable of intervening in the pain processing system, but passive approaches have been little investigated. Among them, little is known about the effect of ischemic preconditioning (IPC) for pain management and its impact on conditioned pain modulation (CPM) and cardiac autonomic control. There is no evidence that IPC causes systemic hypoalgesia and increased vagal modulation, so this provides a rationale for study. Objectives: To analyze the acute effect of IPC on local pain, CPM and cardiac autonomic control in women with knee OA and observe whether there is a correlation between them. Methods: Double-blind, placebo-controlled, randomized clinical trial. Participants will be divided into IPC or placebo groups. Outcomes evaluated: CPM and cardiac autonomic modulation. Comparisons will be performed using Generalized Mixed Linear Models fitted to the data. For correlation, the Pearson or Spearman correlation test will be used according to the normality of the data. All analyzes will assume a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis for uni or bilateral OA of the tibiofemoral joint (grade II or superior Kellgren-Lawrence radiographic changes);
* Not having systemic rheumatic diseases such as fibromyalgia, rheumatoid arthritis, systemic lupus erythematosus;
* Not having total knee arthroplasty, knee ligament injury, history of knee surgery;
* Not having heart disease, congestive heart failure, or a history of acute myocardial infarction (except those with hypertension);
* Not having diagnosis of neurological, metabolic, endocrine disorder, respiratory disease;
* Not being an alcoholic or smoker;
* Not use drugs that influence cardiac autonomic modulation (beta-blocker);
* Not having one or more predisposing risk factors for thromboembolism.

Exclusion Criteria:

* Use anti-inflammatory drugs or analgesics 24 hours before the test;
* Perform physical activity;
* Consume alcohol;
* Perform therapeutic treatments for pain relief;
* Errors in capturing the RR intervals;
* Want to leave the study.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with knee OA, aged 45 years or less and younger than 80 years.
Enrollment: 44 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Conditioned Pain Modulation | Change from baseline after intervention.
  Conditioned pain modulation is a dynamic measure capable of evaluating endogenous pain inhibition using a "pain-by-pain inhibition" model in which pain in a local area (test stimulus) is inhibited by a second concomitant pain (pain stimulus) conditioning). In this study, the test stimulus will be performed through the pressure pain threshold using algometer and the conditioning stimulus will be performed by immersing the hand in cold water, using the cold pressor test - CPT.
Cardiac Autonomic Modulation | Change from baseline after intervention.
  The assessment of cardiac autonomic modulation will be performed using HRV through the capture of heart rate beat to beat (RR intervals) using a heart rate monitor (Polar Electro Oy, Kempele, Finland - model V800) which is a validated equipment.

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Biral TM, de Souza Cavina AP, Junior EP, Filho CATT, Vanderlei FM. Effects of remote ischemic conditioning on conditioned pain modulation and cardiac autonomic modulation in women with knee osteoarthritis: placebo-controlled randomized clinical trial protocol. Trials. 2023 Aug 7;24(1):502. doi: 10.1186/s13063-023-07527-2. PMID 37550703